CLINICAL TRIAL: NCT01792947
Title: Percutaneous Electroneurostimulation of Dermatome T6 for Appetite Reduction and Weight Loss in Morbidly Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Professor, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGUE2013-1
Record Dates: First submitted 2013-02-10; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Appetite Reduction; Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet (Active Comparator): Diet 1200 Kcal during 3 months
  Interventions: Behavioral: Diet 1200 Kcal
- PENS associated to diet (Experimental): Percutaneous electroneurostimulation of dermatome T6 associated to diet 1200 Kcal
  Interventions: Procedure: Percutaneous electroneurostimulation of dermatome T6; Behavioral: Diet 1200 Kcal

INTERVENTIONS:
Procedure: Percutaneous electroneurostimulation of dermatome T6 — The patients underwent a percutaneous electroneurostimulation of dermatome T6 during 30 minutes, every week during 12 weeks. This intervention was associated to a diet 1200 Kcal
  Arms: PENS associated to diet
Behavioral: Diet 1200 Kcal — The patients assigned to this group must follow a 1200 Kcal diet during months

SUMMARY:
Based on the creation of a somato-autonomic reflex, the stimulation of sensory nerve terminals located in dermatome T6 may cause a reflex, whose efferent pathways end in vagal nerve branches stimulating the gastric wall, similarly to the gastric pacemaker.

The aim of this study was to evaluate the effect of percutaneous electroneurostimulation (PENS) of T6 dermatome on appetite, weight loss and dietary compliance.

ELIGIBILITY:
Inclusion Criteria:

* patients candidates to bariatric surgery
* BMI > 40 Kg/m2 or a BMI > 35 Kg/m2 with comorbidities associated to the obesity status
* Failure of dietary treatment.

Exclusion Criteria:

* untreated endocrine disease causing obesity
* serious psychiatric illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Appetite reduction | 3 months
  The appetite reduction will be measured asking the patient to quantify the appetite sensation according to a visula analogic scale, ranged from 0 (absence of appetite) to 10 (incontrolable appetite). Appetite will be measured before the beginning of the treatment and after finishing it (after 12 weeks of treatment).

SECONDARY OUTCOMES:
Weight loss | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ruiz-Tovar, MD, PhD, Principal Investigator — General University Hospital Elche
Locations (1):
- Hospital general Universitario de Elche, Elche, Alicante, Spain

REFERENCES:
- [Derived] Ruiz-Tovar J, Oller I, Diez M, Zubiaga L, Arroyo A, Calpena R. Percutaneous electrical neurostimulation of dermatome T6 for appetite reduction and weight loss in morbidly obese patients. Obes Surg. 2014 Feb;24(2):205-11. doi: 10.1007/s11695-013-1091-z. PMID 24122698